CLINICAL TRIAL: NCT06501066
Title: A Two-part, Phase I/II, Randomized, Single-blind Study to Evaluate the Efficacy and Safety of UMC119-06-05 in Older Adults With Pre-frailty & Frailty
Brief Title: Mesenchymal Stem Cells for Frailty Syndrome
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Meribank Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: UMC119-06-05-FS-12
Record Dates: First submitted 2024-06-18; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Pathologic Processes
Keywords: Frailty; aging; mesenchymal stem cells
MeSH Terms: conditions — Pathologic Processes; Frailty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase I Treatment Arm (Experimental): umbilical cord mesenchymal stem cells, 100×10^6 cells/subject, single treatment by intravenous infusion in phase I.
  Interventions: Biological: umbilical cord mesenchymal stem cells
- Phase II Treatment Arm (Experimental): umbilical cord mesenchymal stem cells, 100×10^6 cells/subject, single treatment by intravenous infusion in phase II.
  Interventions: Biological: umbilical cord mesenchymal stem cells
- Phase II Placebo Arm (Placebo Comparator): Peripheral IV infusion of placebo at baseline.
  Interventions: Biological: umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: umbilical cord mesenchymal stem cells — Patients assigned to UC-MSC administration groups will receive one administrations

SUMMARY:
This Phase I/II study is designed to evaluate the efficacy and safety of UMC119-06-05, an allogeneic umbilical cord mesenchymal stem cells, in older adults with frailty syndrome. This study will also seek to determine the long-term safety and clinical outcomes of UMC119-06-05 in subjects with frailty syndrome, which will provide information for subsequent clinical trials with UMC119-06-05.

DETAILED DESCRIPTION:
Frailty is a disorder of several inter-related physiological systems, including genetic and environmental factors in combination with epigenetic mechanisms, which regulate the differential expression of genes in cells and could be especially important in ageing. Frailty syndrome characterized by a progressive decline in health and clinical symptoms of exhaustion, weight loss, a feeling of slowing down, and a decrease in functional capacity. Current interventions focus on interdisciplinary approaches which include nutritional supplementation, physical exercise, and cognitive intervention. The lack of standardized treatment of the disease resulted in the increasing number of elders diagnosed with frailty. Therefore, development of new therapeutic modalities to improve the clinical outcomes and prognosis of frailty syndrome in adult patients is of urgent need. Recently, preclinical and clinical studies support a cell-based, regenerative treatment strategy i.e., allogenic umbilical cord mesenchymal stem cell therapy may represent a novel therapy for aging frailty. This clinical trial is a phase I/II study. Phase I is an open-label study and all eligible subjects will receive a single-dose IV infusion of UMC119-06-05. Phase II study is a randomized, placebo-controlled, single-blind study and half of eligible subjects will receive a single-dose IV infusion of UMC119-06-05, the others will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for enrollment in the study only if they meet ALL of the following criteria:

1. Subjects of age ≥ 65 years old at screening.
2. Subjects show signs of frailty as assessed by CHS frailty Scores ≥ 1 at screening.
3. Subjects with body weight between 40 kg to 90 kg.
4. Subjects have received standard of care treatment (including exercise and nutritional supplementation) for FS for at least 30 days prior to the study.
5. Subject is willing to provide written informed consent to participate in the study after reading the informed consent form and the information provided.

Exclusion Criteria:

Subjects will be eligible for enrollment in the study only if they meet NONE of the following criteria:

1. Subjects unwilling or unable to perform any of the assessments required by endpoint analysis.
2. Subjects who have a significant comorbid medical condition(s), as judged by the investigator, including, but not limited to:

   1. Confirmed diagnosis of disabling neurologic disorder, including but not limited to Parkinson's disease, Amyotrophic lateral sclerosis, Stroke, or dementia, that significantly impact the assessments for endpoint analysis;
   2. Severe kidney disease requiring hemodialysis or peritoneal dialysis;
   3. Advanced liver disease such as hepatitis or liver cirrhosis;
   4. Severe congestive heart failure (New York Heart Association [NYHA] class 3 and 4);
   5. Autoimmune disease (rheumatoid arthritis, psoriasis/psoriatic arthritis, multiple sclerosis, systemic lupus erythematosus, etc.);
   6. Hearing or visual impairment that significantly impact the assessments for endpoint analysis;
   7. Pulmonary dysfunction requiring steroid therapy or O2 supplementation
   8. Uncontrolled metabolic diseases including type II diabetes mellitus (hemoglobin A1c [HbA1c] > 8.5%)
3. Subjects carry history of malignancy of any organ system (other than curatively treated localized basal or squamous cell carcinoma of the skin, cervical carcinoma in situ) within 5 years prior to the screening visit.
4. Subjects using chronic high dose of steroid (> 5 mg prednisolone or equivalent), immunosuppressant therapy, or TNF-α antagonists.
5. Subjects with human immunodeficiency virus (HIV), active hepatitis B virus (HBV) or hepatitis C virus (HCV) infections.
6. Subjects with known allergy or hypersensitivity to any component of the formulation (normal saline, human serum albumin, or dimethyl sulfoxide).
7. Subjects who have participated in another clinical study of new investigational therapies within 3 months before the study drug administration.
8. Subjects who have received any other stem cell therapy within 12 months before the study drug administration.
9. Subjects have a history of moderate to severe substance use disorder (including alcohol, cannabis, hallucinogens, inhalants, opioids, sedatives/hypnotics/anxiolytics, and stimulants [e.g., amphetamine-type substance, cocaine]) based on Diagnostic and Statistical Manual of Mental Disorders (DSM-5) within the past 3 years.
10. Subjects who have any hospitalization record within one month before the study drug administration (except for the scheduled admission in this study, if required).
11. Subjects who have dramatic change in their standard of care treatment (including exercise and nutritional supplements) for improvement of frailty within one month prior to study treatment, as judged by the investigator.
12. Any other condition that, in the opinion of the investigator, may compromise the safety or compliance of the patient or preclude successful completion of the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs)/ Serious Adverse Events (SAEs). | Up to 12 months through study
  Phase I : Incidence of any treatment-emergent serious adverse events (SAE), defined as the composite of: death, non-fatal pulmonary embolism, stroke, hospitalization for worsening dyspnea and clinically significant laboratory test abnormalities.
Incidence of withdrawals due to adverse events | Up to 12 months through study
  Phase I: Incidence of any treatment-emergent serious adverse events (SAE), defined as the composite of: death, non-fatal pulmonary embolism, stroke, hospitalization for worsening dyspnea and clinically significant laboratory test abnormalities.
vital signs | Up to 12 months through study
  Phase I: change in vital signs
physical examination | Up to 12 months through study
  Phase I: change in physical examination
clinical laboratory test results | Up to 12 months through study
  Phase I: change in clinical laboratory test results
electrocardiogram | Up to 12 months through study
  Phase I: change in electrocardiogram

SECONDARY OUTCOMES:
Mean change from baseline in frailty status (Cardiovascular Health Study [CHS] frailty score | change from baseline to Day 91, Day 181, and Day 361
  CHS scale consists of five components-unintentional weight loss, exhaustion, low activity, weakness, and slowness
Mean change from baseline in grip strength | change from baseline to Day 91, Day 181, and Day 361
  Hand grip strength as assessed by a dynamometer. Grip strength is recorded (in mmHg) three times for each hand.
Mean change from baseline in chair-stand test | change from baseline to Day 91, Day 181, and Day 361
  a subject is able to transfer from a seated to a standing position and back to sitting five times
Mean change from baseline in muscle mass and bone density | change from baseline to Day 91, Day 181, and Day 361
  muscle mass and bone density will be measured using DXA
Mean change from baseline in quality of life measured by change in SF-12 | change from baseline to Day 91, Day 181, and Day 361
  a quality of life measure

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei